CLINICAL TRIAL: NCT04287881
Title: Investigation the Incidence of Methylenetetrahydrofolate Reductase Deficiency in Ischemic Cerebrovascular Diseases Presenting With Epileptic Seizures in Adults
Brief Title: Methylenetetrahydrofolate Reductase Deficiency in Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Nur Orhon, Principal Investigator, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: İstanbulMUZEYNEP2
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Hyperhomocysteinemia, Thrombotic, Cbs-Related; Ischemic Stroke; Epilepsy
Keywords: Methylenetetrahydrofolate reductase (MTHFR) deficiency; Ischemic Stroke; Epileptic seizures; Adult patients
MeSH Terms: conditions — Hyperhomocysteinemia; Ischemic Stroke; Epilepsy; Seizures | interventions — Methylenetetrahydrofolate Reductase (NADPH2)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients who have epileptic seizures (Other): Patients with adult-onset epileptic seizures and diagnosed ischemic stroke.
  Interventions: Genetic: Methylenetetrahydrofolate reductase (MTHFR) deficiency

INTERVENTIONS:
Genetic: Methylenetetrahydrofolate reductase (MTHFR) deficiency — To investigate the incidence of MTHFR deficiency in patients with adult-onset epileptic seizures and diagnosed ischemic stroke

SUMMARY:
Adult onset epileptic seizures is rare and often associated with metabolic disorders, drugs and intracranial pathologies such as ischemia, hemorrhage or space-occupying lesions. Methylenetetrahydrofolate reductase (MTHFR) deficiency is one of the reasons that cause epileptic seizures in adults and can be ignored. MTHFR deficiency is an autosomal recessive disorder that results in hyperhomocysteinemia and causes a predisposition to venous and arterial thrombosis. The incidence of the polymorphism is around 40% in some countries. The aim of the retrospective study is to investigate the incidence of MTHFR deficiency in patients with adult-onset epileptic seizures.

DETAILED DESCRIPTION:
Epileptic seizures that begin in adulthood seriously affect patients, their relatives and the society in which they live financially and psychologically. The etiology of epileptic seizures starting at adult age includes head trauma, central nervous system infections, intracranial lesions, cerebrovascular events, metabolic diseases and drugs. While the causes of childhood epileptic seizures are generally considered idiopathic, adult-onset epileptic seizures are almost always due to a pathological process. Epileptic seizures in adults may be a symptom of ischemic stroke. MTHFR deficiency is associated with raised homocysteine concentration in the body and increased risk of stroke (1). Studies have demonstrated that hyperhomocysteinemia is an independent risk factor for stroke (2).

MTHFR is the key enzyme in remethylation of homocysteine to methionine. MTHFR deficiency is an autosomal-recessive disease characterized by high homocysteine and low or normal methionine. MTHFR deficiency can cause vascular thrombosis in adults at early age; increased osteoporosis in elderly people; deep vein thrombosis, abortus during pregnancy; and infertility in adult males. In children, it is associated with intrauterine growth retardation, congenital heart diseases, neural tube defects, chromosome anomalies and hematologic tumors. In any age group, it might cause convulsions, increased thrombosis risk with some anticonvulsants and with the use of nitrogen protoxide in surgeries, and neuromotor retardation (3).

The aim of this retrospective study is to investigate the incidence of MTHFR deficiency in patients presenting with adult-onset epileptic seizures and diagnosed as ischemic cerebrovascular disease as a result of diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* The patients with adult-onset epileptic seizures and diagnosed ischemic stroke in 3 years period.

Exclusion Criteria:

* Pediatric patients with epileptic seizures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Methylenetetrahydrofolate reductase (MTHFR) deficiency | Up to 6 weeks
  The incidence of methylenetetrahydrofolate reductase (MTHFR) deficiency in ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP ORHON, MD, Principal Investigator — Istanbul Medeniyet University
Locations (2):
- Turkey (Türkiye) (2):
  - Zeynep Orhon, Istanbul
  - Istanbul MU Goztepe Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No